CLINICAL TRIAL: NCT03369184
Title: Elective Percutaneous Coronary Intervention With or Without Supplemental OXYgen and Evaluation of Effects on Coronary Microcirculation Using the Index of Microcirculatory Resistance
Brief Title: Elective Percutaneous Coronary Intervention With or Without Supplemental OXYgen
Acronym: EPOXY-IMR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Nils Witt, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-10.1
Record Dates: First submitted 2017-11-28; First posted 2017-12-11 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary flow; Coronary vascular resistance; Supplemental oxygen
MeSH Terms: conditions — Coronary Artery Disease | interventions — nitrox; Particulate Matter

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patients are randomized in a double blinded fashion by a designated study nurse (simple envelope randomization) to either supplemental oxygen 6l/min delivered by an open face mask (Oxymask®) or ambient air (sham placement of Oxymask®). Neither the patient, nor the performing physician will be aware of the randomization status. Peripheral oxygen saturation will be disclosed only to the nurse responsible for randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supplemental oxygen (Experimental): Inhalation of oxygen 6 L/min through an open face mask
  Interventions: Drug: Oxygen gas
- Ambient air (Sham Comparator): Breathing ambient air through an open face mask
  Interventions: Other: Ambient air

INTERVENTIONS:
Drug: Oxygen gas — The intervention is administered as previously described. The duration of intervention is 10 minutes.
  Arms: Supplemental oxygen
Other: Ambient air — Administered similarly to treatment arm, via an open face mask and during 10 minutes
  Arms: Ambient air

SUMMARY:
Supplemental oxygen is frequently used in patients admitted to hospital due to ischemic heart disease. In the setting of suspected myocardial infarction, clinical practice guidelines advocate the use of supplementary oxygen even in patients with normal levels of peripheral oxygen saturation. The theoretical basis for this practice is that an increase in blood oxygen content may limit ischemia and final myocardial damage and subsequent infarct size. However, although some experimental laboratory data and small studies in humans have supported the use of supplemental oxygen in patients with coronary artery disease, contradicting evidence suggests possible harmful effects, mainly through mechanisms involving coronary vasoconstriction and reduction of myocardial perfusion (hyperoxemic coronary vasoconstriction).

In the EPOXY-IMR trial, the investigators aim to further explore possible detrimental effects from routine use of supplemental oxygen on the coronary circulation with special focus on the small vessels referred to as the coronary microcirculation.

DETAILED DESCRIPTION:
Aim:

The aim of the EPOXY-IMR trial is to evaluate the effect of supplemental oxygen on coronary circulation in the setting of elective coronary angiography and percutaneous coronary intervention (PCI). To achieve this, different functional parameters such as the index of microcirculatory resistance (IMR), fractional flow reserve (FFR) and coronary flow reserve (CFR) will be obtained and serial biomarkers (cardiac troponin) will be analyzed.

Background:

Coronary artery disease (CAD) based on arteriosclerotic narrowing of the coronary blood vessels is the most common cause of death in the western world. To determine the severity of the disease in symptomatic patients and guide optimal therapy, coronary angiography is frequently performed. Simplified, three outcomes can be found:

1. No or mild evidence of CAD leading to continuous medical therapy.
2. Severe disease demanding revascularization therapy done by either percutaneous coronary intervention (PCI), where most commonly balloon dilatation followed by placement of a metal stent in the coronary vessel is performed, or coronary artery bypass grafting (CABG).
3. In patients with moderate disease further functional testing is required to assess the gravity of the narrowing. This can be achieved by placing a pressure sensor equipped guide wire to the diseased artery comparing blood pressure proximal and distal to the stenosis during hyperemia, known as Fractional Flow Reserve (FFR). Although based on pressure recordings, FFR is a highly accurate measure of the flow limitation of a given stenosis. A common cut-off value of 0,8 is used where a lower value mandates therapy as in patients with severe disease.

Further information regarding the coronary circulation can be obtained by calculation of coronary flow reserve (CFR) and the index of microcirculatory resistance (IMR), the former representing a measure of the flow situation in the complete coronary arterial system, the latter more specifically the vascular resistance in the microcirculatory compartment. These indices are based on thermodilution measurements using a temperature sensor also located in the above mentioned pressure sensor equipped guide wire.

Supplemental oxygen is frequently used all over the world in patients hospitalized with suspected coronary artery disease (CAD) irrespective of oxygen levels in the blood. Scientifically, only experimental laboratory data and small studies in humans have supported this practice.

In contrast, mounting evidence suggests possible harmful effects of supplemental oxygen by causing a decrease in cardiac function, especially through mechanisms of narrowing of the coronary arteries due high oxygen levels in the blood (hyperoxemic coronary vasoconstriction). Clinically, epicardial coronary vasoconstriction mediated by oxygen therapy may result in underestimation of vessel size during percutaneous coronary intervention (PCI), possibly increasing the risk of subsequent complications such as stent thrombosis and in-stent restenosis. Furthermore, vasoconstriction in the microcirculatory compartment may result in increased periprocedural myocardial injury as a result of microvascular obstruction from plaque related and thrombotic material.

In the EPOXY-IMR trial, the investigators aim to analyze possible detrimental effects of supplemental oxygen in patients undergoing coronary angiography and intracoronary pressure/flow measurements due to angiographically intermediate coronary lesions and with special focus on the circulation of the small vessels (microvascular function).

Design:

EPOXY-IMR is a single centre, interventional, double-blinded, randomized, controlled trial aiming to recruit 40 patients in the treatment group (cohort A, patients in whom PCI is performed) and 25 patients in the non-intervention group (cohort B, patients in whom PCI is deferred on the basis of a non-significant FFR-value).

Materials and methods:

Patients with suspected coronary artery disease (CAD) scheduled for elective coronary angiography and normal oxygen saturation (≥90% on pulse oximeter) are asked to participate in the trial in good time prior to the exam. After written informed consent standard diagnostic coronary angiography is performed. If coronary stenosis of moderate degree is found in the larger arteries (40-90% diameter stenosis), further functional evaluation is mandated to determine if the stenosis impedes coronary blood flow significantly. According to clinical routine, this is achieved by placing a pressure wire in the diseased vessel passing the narrowed section, obtaining data on coronary blood pressure proximal and distal to the stenosis and inducing hyperemia with adenosine infusion for determination of FFR. Using thermodilution with intracoronary bolus injections of room temperature saline, data for calculation of the index of microcirculatory resistance (IMR) and coronary flow reserve (CFR) will be obtained.

Those patients with FFR <0,8 indicative of restricted blood flow to the heart muscle mandating further treatment by PCI, form cohort A. Patients with FFR >0,8 make up cohort B.

Thereafter, the patients are randomized in a double blinded fashion by a designated study nurse to either supplemental oxygen 6l/min delivered by an open face mask (Oxymask®) or ambient air (sham placement of Oxymask®).

Cohort A: After 10 minutes inhalation of oxygen/ambient air, FFR, CFR and IMR are re-measured followed by PCI according to clinical routine. Finally, post PCI measurements of IMR, FFR and CFR are performed. Troponin levels are obtained at baseline, 4 hours and 12-24 hours post PCI. An arterial blood gas sample is drawn just before PCI. During PCI, coronary pressure distal to the lesion is recorded during balloon inflation, allowing for recording of wedge pressure which is required for correct calculation of flow- and resistance indices in a significantly stenosed vessel.

Cohort B: After 10 minutes inhalation of oxygen/ambient air, FFR, CFR and IMR are re-measured

Hypothesis:

* Supplemental oxygen reduces coronary blood flow and increases microcirculatory resistance
* Supplemental oxygen increases microcirculatory resistance leading to increased procedure related myocardial damage

Primary endpoint is the effect of supplemental oxygen on IMR. Secondary endpoints will furthermore evaluate effects on CFR, FFR and serial cardiac troponin.

Conclusion:

To date, there is limited and conflicting evidence supporting the routine administration of supplemental oxygen in patients with coronary artery disease. The EPOXY-IMR trial is designed to explore the effects of supplemental oxygen on coronary blood flow and microvascular resistance as potential mediators of detrimental clinical effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age, AND
* Undergoing elective coronary angiography due to suspected stabile coronary artery disease
* Evidence of moderate (40%-79%) stenosis, requiring further routine assessment with FFR.
* Informed consent

Exclusion Criteria:

* Acute coronary syndrome or myocardial infarction within 7 days
* Hypoxia with oxygen saturation measured on pulse oximeter < 90% with the patient breathing air
* Left ventricular hypertrophy on echocardiography (septum >13mm)
* Asthma (not COPD)
* Advanced AV-block without pacemaker in situ
* Altered conscious state/inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Index of Microcirculatory Resistance (IMR) | Change from baseline to 1 hour
  Measure of microvascular resistance. Intracoronary pressure- and flow-based measurements derived from thermodilution recordings.

SECONDARY OUTCOMES:
Coronary Flow Reserve (CFR) | Change from baseline to 1 hour
  Flow-related index based om thermodilution measurements
High sensitive troponin | Measured at baseline, after 4, 12 and 24 hours.
  Cardiac biomarker and a measure of periprocedural myocardial damage

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm South General Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Santos-Pardo I, Alstrom P, Witt N. Index of Microcirculatory Resistance Measured during Intracoronary Adenosine-Induced Hyperemia. J Interv Cardiol. 2020 May 12;2020:4829647. doi: 10.1155/2020/4829647. eCollection 2020. PMID 32508541